CLINICAL TRIAL: NCT02040480
Title: A Single Center, Randomized, Open-Label, Sequential, Single Dose, 3-Period Crossover Study to Evaluate the Bioavailability and Food Effect of a Gelatin Formulation and Immediate Release Tablet Formulation of Afuresertib, an AKT Inhibitor, in Normal Healthy Volunteers
Brief Title: Bioavailability and Food Effect Study of Gelatin Formulation and Immediate Release Tablet Formulation of Afuresertib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201039
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Cancer
Keywords: bioavailability; food effect; formulation; GSK2110183; afuresertib; AKT inhibitor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1 (Experimental): Participants will receive treatment in following sequence in each of the three study periods (one treatment per period): ABC
  Interventions: Drug: GSK2110183 Gelatin Capsule; Drug: GSK2110183 IR Tablet
- Sequence 2 (Experimental): Participants will receive treatment in following sequence in each of the three study periods (one treatment per period): ACB
  Interventions: Drug: GSK2110183 Gelatin Capsule; Drug: GSK2110183 IR Tablet
- Sequence 3 (Experimental): Participants will receive treatment in following sequence in each of the three study periods (one treatment per period): BAC
  Interventions: Drug: GSK2110183 Gelatin Capsule; Drug: GSK2110183 IR Tablet
- Sequence 4 (Experimental): Participants will receive treatment in following sequence in each of the three study periods (one treatment per period): BCA
  Interventions: Drug: GSK2110183 Gelatin Capsule; Drug: GSK2110183 IR Tablet
- Sequence 5 (Experimental): Participants will receive treatment in following sequence in each of the three study periods (one treatment per period): CAB
  Interventions: Drug: GSK2110183 Gelatin Capsule; Drug: GSK2110183 IR Tablet
- Sequence 6 (Experimental): Participants will receive treatment in following sequence in each of the three study periods (one treatment per period): CBA
  Interventions: Drug: GSK2110183 Gelatin Capsule; Drug: GSK2110183 IR Tablet

INTERVENTIONS:
Drug: GSK2110183 Gelatin Capsule — White opaque hard gelatin capsule with a unit dose strength of 25 milligrams (mg) for oral administration
Drug: GSK2110183 IR Tablet — White round biconvex film coated IR tablet with a unit dose strength of 25 mg for oral administration

SUMMARY:
This study is being conducted to measure the relative bioavailability of the original gelatin capsule formulation and a new formulation, immediate release (IR) tablet of Afuresertib (GSK2110183). The study will be composed of Screening, Treatment, and Follow-up Periods. A subject's total time involved in the study will be approximately 9 weeks. The study will enroll approximately 18 healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Provided signed written informed consent
* Healthy Male or female between 18 and 40 years of age inclusive, at the time the informed consent is obtained.
* Body weight >=50 kilograms (kg) and body mass index (BMI) of >=18 and <= 32 kg/meter square (m^2).
* A female subject is eligible to participate if she is of (A) Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy or postmenopausal defined as 12 months of spontaneous amenorrhea (B) Child-bearing potential with negative pregnancy test as determined by serum human chorionic gonadotropin (hCG) test at Screening and prior to dosing, AND: agrees to use one of the acceptable contraception methods
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods.
* Alanine aminotransferase, alkaline phosphatase and bilirubin <=1.5xupper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Based on single or averaged QT interval corrected (QTc) values of triplicate ECGs obtained over a brief recording period: QTcB <450 millisecond (msec); or QTcB <480 msec in subjects with Bundle Branch Block.
* Able to swallow and retain orally administered study treatment and does not have any clinically significant gastrointestinal (GI) abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach and/or bowels.

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of gastroesophageal reflux disease, dyspepsia, peptic ulcer disease, gastrointestinal (GI) bleeding, GI surgery that could affect motility.
* History of atrial arrhythmias
* History of regular alcohol consumption within 6 months of the study defined as:

An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 10 grams (g) of alcohol: 270 mL of full strength beer (4.8%), 375 mL of mid strength beer (3.5%), 470 mL of light beer (2.7%), 250 mL pre-mix full strength spirit (5%), 100mL of wine (13.5%) and 30 mL of spirit (40%).

* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or GSK Medical Monitor, contraindicates their participation
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of Screening.
* Smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* A positive drug/alcohol screen at Screening or upon check-in to the clinic on Day -1 of each Dosing Period.
* A positive test for human immuno virus (HIV) antibody.
* Pregnant females as determined by positive serum hCG test at Screening or prior to dosing.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Lactating females.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures.
* Any prohibited medications or recent consumption of citrus products.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-02-05 (Actual); Primary Completion 2014-04-04 (Actual); Study Completion 2014-04-04 (Actual)

PRIMARY OUTCOMES:
Composite of pharmacokinetic (PK) parameters to determine relative bioavailability of afuresertib after administering it as a single dose in an original gelatin capsule in the fasted state and in a newly formulated IR tablet in the fed and fasted state. | PK Samples will be collected Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 120, and 168 hours post-dose
  PK parameters include: area under the plasma concentration-time curve from time zero to infinity (AUC [0-infinity]), area under the plasma concentration time curve from time zero to last time of quantifiable concentration (AUC [0-t]), maximum observed plasma concentration (Cmax), and time to Cmax (tmax).

SECONDARY OUTCOMES:
Number of subjects with adverse events (AEs). | Up to 9 weeks
  AEs will be collected from the start of Study Treatment and until the Follow-up contact.
Clinical laboratory parameter assessment as a measure of safety and tolerability | Up to 9 weeks
  Laboratory parameters include: hematology, clinical chemistry and urinalysis.
Concomitant medications review as a measure of safety and tolerability | Up to 9 weeks
Electrocardiogram (ECGs) measurement as a measure of safety and tolerability | Up to 9 weeks
  Triplicate 12-lead ECGs will be collected at Screening; in each Dosing Period on Day 1 and Day 3 of Dosing Period; and at Follow-up.
Vital sign measurement as a measure of safety and tolerability | Up to 9 weeks
  Vital sign measurements will include systolic and diastolic blood pressure and pulse rate.
Composite of PK parameter following single dose administration of IR tablet in fasted state | PK Samples will be collected Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 120, and 168 hours post-dose
  PK parameters include: AUC (0 - infinity), AUC (0 - t), Cmax, and tmax.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

REFERENCES:
- See also: Results for study 201039 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/201039?search=study&search_terms=201039#rs